CLINICAL TRIAL: NCT01507428
Title: Randomized Phase II Trial of Individualized Adaptive Radiotherapy Using During-Treatment FDG-PET/CT and Modern Technology in Locally Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Study of Positron Emission Tomography and Computed Tomography in Guiding Radiation Therapy in Patients With Stage III Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-00107; NCI-2012-00107 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000721619; RTOG-1106/ACRIN-6697; RTOG-1106 (Other: NRG Oncology); RTOG-1106 (Other: CTEP); U10CA180868 (NIH); U10CA021661 (NIH)
Record Dates: First submitted 2012-01-05; First posted 2012-01-10 (Estimated); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Stage III Lung Non-Small Cell Cancer AJCC v7; Stage IIIA Lung Non-Small Cell Cancer AJCC v7; Stage IIIB Lung Non-Small Cell Cancer AJCC v7
MeSH Terms: interventions — fluoromisonidazole; Carboplatin; Radiation; Fluorodeoxyglucose F18; Paclitaxel; Taxes; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (standard chemoradiotherapy) (Active Comparator): Patients undergo radiotherapy QD 5 days a week for 30 fractions. Patients also receive paclitaxel IV over 1 hour and carboplatin IV over 30 minutes once weekly for 6 weeks. Patients undergo FDG-PET/CT imaging between fractions 18 and 19.
  Interventions: Drug: 18F-Fluoromisonidazole; Drug: Carboplatin; Procedure: Computed Tomography; Radiation: External Beam Radiation Therapy; Drug: Fludeoxyglucose F-18; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Procedure: Positron Emission Tomography
- Arm II (experimental chemoradiotherapy) (Experimental): Patients undergo an individualized dose of image-guided radiotherapy QD 5 days a week for 30 fractions and undergo 18 F FDG-PET/CT between fractions 18 and 19. Based on the scan results, patients undergo individualized adaptive radiotherapy for the final 9 fractions. Patients also receive paclitaxel and carboplatin as in Arm I.
  Interventions: Drug: 18F-Fluoromisonidazole; Drug: Carboplatin; Procedure: Computed Tomography; Drug: Fludeoxyglucose F-18; Radiation: Image-Guided Adaptive Radiation Therapy; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Procedure: Positron Emission Tomography

INTERVENTIONS:
Drug: 18F-Fluoromisonidazole — Undergo FMISO PET/CT (Correlative studies)
  Other Names: 18F-MISO; 18F-Misonidazole; FMISO
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Procedure: Computed Tomography — Undergo FDG PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Procedure: Computed Tomography — Undergo FMISO PET/CT (Correlative studies)
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Radiation: External Beam Radiation Therapy — Undergo radiotherapy
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam
  Arms: Arm I (standard chemoradiotherapy)
Drug: Fludeoxyglucose F-18 — Undergo FDG PET/CT
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Radiation: Image-Guided Adaptive Radiation Therapy — Undergo individualized adaptive radiotherapy
  Other Names: IGART
  Arms: Arm II (experimental chemoradiotherapy)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Procedure: Positron Emission Tomography — Undergo FDG PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Procedure: Positron Emission Tomography — Undergo FMISO PET/CT (Correlative studies)
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This randomized phase II trial studies how well positron emission tomography (PET)/computed tomography (CT)-guided radiation therapy works compared to standard radiation therapy in treating patients with stage III non-small cell lung cancer. Radiation therapy uses high-energy x-rays to kill tumor cells. Using imaging procedures, such as PET and CT scans, to guide the radiation therapy, may help doctors deliver higher doses directly to the tumor and cause less damage to healthy tissue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether tumor dose can be escalated to improve the freedom from local-regional progression-free (LRPF) rate at 2 years when an individualized adaptive radiation treatment (RT) plan is applied by the use of a fludeoxyglucose F 18 (FDG)-positron emission tomography (PET)/computed tomography (CT) scan acquired during the course of fractionated RT in patients with inoperable stage III non-small cell lung cancer (NSCLC). (National Surgical Adjuvant Breast and Bowel Project [NSABP], Radiation Therapy Oncology Group [RTOG], Gynecologic Oncology Group [GOG] [NRG] Oncology) II. To determine whether the relative change in standard uptake value (SUV) peak from the baseline to the during-treatment FDG-PET/CT, defined as (during-treatment SUVpeak - baseline SUVpeak)/baseline SUV peak x 100%, can predict the LRPF rate with a 2-year follow up. (Eastern Cooperative Oncology Group [ECOG]-American College of Radiology Imaging Network [ACRIN])

SECONDARY OBJECTIVES:

I. To determine whether an individualized dose escalation improves overall survival (OS), progression-free survival (PFS), lung cancer cause-specific survival, and delays time to local-regional progression compared to a conventional RT plan. (NRG Oncology) II. To compare the rate of severe (grade 3+ Common Terminology Criteria for Adverse Events [CTCAE], v. 4) radiation-induced lung toxicity (RILT) defined as severe RILT pneumonitis or clinical fibrosis. (NRG Oncology) III. To compare other severe adverse events, including grade 3+ (CTCAE, v. 4) esophagitis or grade 2 pericardial effusions, or any grade cardiac adverse events related to chemoradiation between a PET/CT-guided adaptive approach and a conventional RT plan. (NRG Oncology) IV. To evaluate the association of baseline 18F-fluoromisonidazole (FMISO), a PET/CT imaging agent uptake (tumor-to-blood pool ratio) with LRPF (i.e., the assessment of using baseline FMISO-PET uptake as a prognostic marker). (ECOG-ACRIN) V. To determine if the relative change in SUVpeak from baseline to during-treatment FDG-PET/CT and/or baseline FMISO uptake (tumor-to-blood pool ratio) predicts the differential benefit of the adaptive therapy, i.e., the association of uptake parameters with LRPF rate depending on the assigned treatment thus, assessing if these uptake parameters can be useful in guiding therapies, i.e., predictive markers. (ECOG-ACRIN) VI. To determine if other PET-imaging uptake parameters (SUV peak during-treatment for FDG-PET, maximum SUV, or relative change of maximum SUVs from pre- to during-treatment FDG-PET/CT, change in metabolic tumor volume, FMISO total hypoxic volume, FMISO tumor to mediastinum ratio, EORTC or University of Michigan/Kong's response criteria) will predict OS, LRPF rate, and lung cancer cause-specific (LCS) survival as well as to explore the optimal threshold for differentiating responders from non-responders. (ECOG-ACRIN)

CORRELATIVE SCIENCE OBJECTIVES:

I. To study whether a model of combining current clinical and/or imaging factors with blood markers, including osteopontin (OPN) [for hypoxia marker], carcinoembryonic antigen (CEA) and cytokeratin fragment (CYFRA) 21-1 (for tumor burden), and interleukin (IL)-6 (inflammation) will predict the 2-year LRPF rate and survival better than a current model using clinical factors and radiation dose as well as imaging factors.

II. To determine/validate whether a model of combining mean lung dose (MLD), transforming growth factor beta1 (TGF beta1) and IL-8 will improve the predictive accuracy for clinical significant RILT better comparing to the current model of using MLD alone.

III. To explore, in a preliminary manner, whether proteomic and genomic markers in the blood prior to and during the early course of treatment are associated with tumor response after completion of treatment, LRPF rate, PFS, OS, and pattern of failure and treatment-related adverse events, such as radiation pneumonitis, esophagitis, and pericardial effusion. (exploratory)

OUTLINE:

Prior to treatment, patients undergo fludeoxyglucose F 18 (FDG) positron emission tomography (PET) and computed tomography (CT) scans at baseline and periodically during study. A subset of patients also undergo 18F-fluoromisonidazole PET/CT scan at baseline. Patients are randomized to 1 of 2 treatment arms:

ARM I (standard chemoradiotherapy): Patients undergo radiotherapy once daily (QD) 5 days a week for 30 fractions. Patients also receive paclitaxel intravenously (IV) over 1 hour and carboplatin IV over 30 minutes once weekly for 6 weeks. Patients undergo FDG-PET/CT imaging between fractions 18 and 19.

ARM II (experimental chemoradiotherapy): Patients undergo an individualized dose of image-guided radiotherapy QD 5 days a week for 30 fractions and undergo 18 F FDG-PET/CT between fractions 18 and 19. Based on the scan results, patients undergo individualized adaptive radiotherapy for the final 9 fractions. Patients also receive paclitaxel and carboplatin as in Arm I.

CONSOLIDATION CHEMOTHERAPY: Beginning 4-6 weeks after chemoradiotherapy, patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 1 month, every 3 months for 1 year, every 6 months for 2 years, and then annually for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have FDG-avid (maximum SUV >= 4.0) (from PET scan of any date, any scanner) and histologically or cytologically proven non-small cell lung cancer
* Patients must be clinical American Joint Committee on Cancer (AJCC) stage IIIA or IIIB (AJCC, 7th ed.) with non-operable disease; non-operable disease will be determined by a multi-disciplinary treatment team, involving evaluation by at least 1 thoracic surgeon within 8 weeks prior to registration; Note: For patients who are clearly nonresectable, the case can be determined by the treating radiation oncologist and a medical oncologist, or pulmonologist
* Patients with multiple, ipsilateral pulmonary nodules (T3 or T4) are eligible if a definitive course of daily fractionated radiation therapy (RT) is planned
* History/physical examination, including documentation of weight, within 2 weeks prior to registration
* FDG-PET/CT scan for staging and RT plan within 4 weeks prior to registration
* CT scan or sim CT of chest and upper abdomen (IV contrast is recommended unless medically contraindicated) within 6 weeks prior to registration
* CT scan of the brain (contrast is recommended unless medically contraindicated) or MRI of the brain within 6 weeks prior to registration
* Pulmonary function tests, including diffusion capacity of carbon monoxide (DLCO), within 6 weeks prior to registration; patients must have forced expiratory volume in 1 second (FEV1) >= 1.2 Liter or >= 50% predicted without bronchodilator
* Zubrod performance status 0-1
* Able to tolerate PET/CT imaging required to be performed at an American College of Radiology (ACR) Imaging Core Laboratory (Lab) qualified facility
* Absolute neutrophil count (ANC) >= 1,500 cells/mm^3 (within 2 weeks prior to registration on study)
* Platelets >= 100,000 cells/mm^3 (within 2 weeks prior to registration on study)
* Hemoglobin (Hgb) >= 10.0 g/dL (note: the use of transfusion or other intervention to achieve Hgb >= 10.0 g/dL is acceptable) (within 2 weeks prior to registration on study)
* Serum creatinine within normal institutional limits or a creatinine clearance >= 60 ml/min within 2 weeks prior to registration
* Negative serum or urine pregnancy test within 3 days prior to registration for women of childbearing potential
* Women of childbearing potential and male participants must agree to use a medically effective means of birth control throughout their participation in the treatment phase of the study
* The patient must provide study-specific informed consent prior to study entry

Exclusion Criteria:

* Patients with any component of small cell lung carcinoma are excluded
* Patients with evidence of a malignant pleural or pericardial effusion are excluded
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years (for example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible)
* Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Severe, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol
  * Acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control (CDC) definition; note, however, that human immunodeficiency virus (HIV) testing is not required for entry into this protocol
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception
* Poorly controlled diabetes (defined as fasting glucose level > 200 mg/dL) despite attempts to improve glucose control by fasting duration and adjustment of medications; patients with diabetes will preferably be scheduled in the morning and instructions for fasting and use of medications will be provided in consultation with the patients' primary physicians
* Patients with T4 disease with radiographic evidence of massive invasion of a large pulmonary artery and tumor causing significant narrowing and destruction of that artery are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2012-02-22 (Actual); Primary Completion 2020-08-17 (Actual); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Local-regional, progression-free (LRPF) rate (National Surgical Adjuvant Breast and Bowel Project [NSABP], Radiation Therapy Oncology Group [RTOG], Gynecologic Oncology Group [GOG] [NRG]) | 2 years
Relative change in standard uptake volume (SUV) peak from the baseline to the during-treatment fludeoxyglucose F 18 (FDG)-positron emission tomography (PET)/computed tomography (CT) to LRPF (ECOG-ACRIN) | Baseline to 2 years

SECONDARY OUTCOMES:
Time to local-regional progression (NRG) | Interval from registration to date of local or regional progression, assessed up to 5 years
Overall survival (OS) (NRG) | Interval from registration to the date of death or censored at the date of data collection, assessed up to 5 years
Progression free survival (PFS) (NRG) | Interval from the date of registration to the date of tumor progression locally, regionally, distantly, or death, whichever occurs first, or censored at the last date of data collection, assessed up to 5 years
Lung cancer cause-specific survival (NRG) | Interval from the date of registration to the date of death directly from lung cancer, or censored at the last date of data collection if still alive, assessed up to 5 years
Radiation-induced lung toxicity (NRG) | Up to 5 years
Incidence of grade 3+ esophagitis or cardiac adverse events related to chemoradiation between a conventional RT plan and a PET/CT-guided adaptive RT plan, as measured by Common Terminology Criteria for Adverse Events, version 4 and 5 (NRG) | Up to 5 years
Baseline 18F-fluoromisonidazole (FMISO) uptake (tumor-to-blood pool ratio) association with LRPF (i.e. the assessment of using baseline FMISO-PET uptake as a prognostic marker) (ECOG-ACRIN) | Baseline
Relative change in SUV peak from the baseline to the during-treatment FDG PET/CT and/or the baseline FMISO uptake (tumor-to-blood pool ratio) prediction of the differential benefit of the adaptive therapy (ECOG-ACRIN) | Baseline to up to 5 years
Change of peak SUVs for FDG from pre- to during-treatment (ECOG-ACRIN) | Baseline to up to 5 years
Max SUV or change of max SUVs for FDG from pre- to during-treatment (ECOG-ACRIN) | Baseline to up to 5 years
Change in metabolic tumor volume (ECOG-ACRIN) | Baseline to up to 5 years
FMISO total hypoxic volume (ECOG-ACRIN) | Up to 5 years
FMISO tumor-to-blood pool ratio (ECOG-ACRIN) | Up to 5 years
Prediction of OS, LRPF, and lung cancer cause-specific survival (ECOG-ACRIN) | Up to 5 years
Optimal threshold for differentiating responders from non-responders (ECOG-ACRIN) | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Ming (Spring) P Kong, Principal Investigator — NRG Oncology
Locations (31):
- United States (29):
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Augusta University Medical Center, Augusta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Sleepy Hollow, Sleepy Hollow, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - McGill University Department of Oncology, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Kong FS, Hu C, Pryma DA, Duan F, Matuszak M, Xiao Y, Ten Haken R, Siegel MJ, Hanna L, Curran WJ, Dunphy M, Gelblum D, Piert M, Jolly S, Robinson CG, Quon A, Loo BW, Srinivas S, Videtic GM, Faria SL, Ferguson C, Dunlap NE, Kundapur V, Paulus R, Siegel BA, Bradley JD, Machtay M. Primary Results of NRG-RTOG1106/ECOG-ACRIN 6697: A Randomized Phase II Trial of Individualized Adaptive (chemo)Radiotherapy Using Midtreatment 18F-Fluorodeoxyglucose Positron Emission Tomography/Computed Tomography in Stage III Non-Small Cell Lung Cancer. J Clin Oncol. 2024 Nov 20;42(33):3935-3946. doi: 10.1200/JCO.24.00022. Epub 2024 Oct 4. PMID 39365957

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/28/NCT01507428/Prot_SAP_000.pdf